CLINICAL TRIAL: NCT05373004
Title: Comparison Between the Efficacy of Sodium-Glucose Co-transporter 2 Inhibitor Therapy Versus Angiotensin-converting Enzyme Inhibitor in the Treatment of Diabetic Kidney Disease
Brief Title: Comparison Between the Efficacy of SGLT2 Inhibitor Therapy Versus ACE Inhibitor in the Treatment of Diabetic Kidney Disease
Acronym: SGLT2i VS ACEi
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Omar Tarek Elfarargi (Other Government)
Responsible Party: Sponsor-Investigator, Omar Tarek Elfarargi, principle investigator, Hamad General Hospital
Organization: Hamad General Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 54520
Record Dates: First submitted 2022-05-05; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Nephropathy Type 2
Keywords: diabetic kidney disease (DKD); SGLT2 inhibitors; ACE inhibitors
MeSH Terms: conditions — Diabetic Nephropathies | interventions — empagliflozin; Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The trial will be double-blinded including both participants and health care providers to minimize the risk of bias. The blinding of outcome adjudicators and data collectors is unlikely to matter since the study outcomes are objective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin 25 mg arm (SGLT2 inhibitor) (Experimental): empagliflozin 10 mg once daily plus a placebo enalapril 10 mg tab, along with conventional antihypertensive (for hypertension patients) & glycemic control therapies (if present). After four weeks, the dose of empagliflozin will be increased to 25 mg once (with Enalapril 20 mg placebo) daily throughout the study for one year.
  Interventions: Drug: Empagliflozin 25 MG
- Enalapril 20 mg arm (ACE inhibitor) (Active Comparator): enalapril 10 mg tab once daily plus a placebo empagliflozin 10 mg tab, along with conventional antihypertensive (for hypertension patients) & glycemic control therapies (if present). After four weeks, the dose of enalapril will be increased to 20 mg once (with Empagliflozin 25 mg placebo) daily throughout the study for one year.
  Interventions: Drug: Enalapril Maleate 20 mg

INTERVENTIONS:
Drug: Empagliflozin 25 MG — It is the experimental drug in this trial. this drug has an approved efficacy in delaying kidney deterioration based on the results of (the EMPA-REG OUTCOME) trial. it is also recommended based on the ADA/EASD 2019 consensus, as the SGLT2 inhibitors are recommended in patients with type 2 diabetes in patients with CKD to prevent the progression of CKD. However, the previous trials where always add it to a patient already on an ACE inhibitor (in most cases). In this trial, it will be compared head to head with the gold standard treatment of CKD which is Enalapril 20 mg (ACE inhibitor).
  Other Names: Jardiance 25 MG
  Arms: Empagliflozin 25 mg arm (SGLT2 inhibitor)
Drug: Enalapril Maleate 20 mg — It is an ACE inhibitor, the active comparator in this trial, and is considered the gold standard for the treatment of diabetic kidney disease.
  Other Names: Renitec 20 MG
  Arms: Enalapril 20 mg arm (ACE inhibitor)

SUMMARY:
Diabetes is the leading cause of chronic kidney disease (CKD) and end-stage kidney disease worldwide. Diabetic kidney disease (DKD) is a clinical diagnosis based upon the presence of reduced glomerular filtration rate (GFR) and/or increased urinary albumin excretion (UACR) in diabetes. The inhibition of the renin-angiotensin system (RAS) has been identified as the cornerstone in the management of DKD for decades. Recently, more evidence supports the use of Sodium-glucose cotransporter 2 inhibitors (SGLT2i) in the treatment of DKD. They were associated with slower progression of renal disease and lower rates of clinically relevant kidney events. Those studies confirmed the SGLT2i efficacy in kidney protection and showed that their addition to angiotensin-converting enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARBS) will be more effective than using ACEi or ARBS alone. It is unclear whether SGLT2i is used as a first-line instead of ACEi or ARB, and to what extent it will be effective in managing DKD compared to the proven effect of ACEi/ARBs alone. This study provides a unique opportunity to address this gap in the literature.

The aim of this study is to compare, head to head, the renal performance of ACEi (standard of care) versus SGLT2 in diabetic patients who have evidence of deteriorating renal function evidenced by either the reduction of e GFR or increased UACR.

Scientific hypotheses:

Null hypothesis:

after one year, the mean change of the e GFR in the enalapril group - Mean change of the e GFR in the empagliflozin group > or = 5 ml/min/1.73m2

Alternative hypothesis:

after one year, the mean change of the e GFR in the enalapril group - Mean change of the e GFR in the empagliflozin group < 5 ml/min/1.73m2

DETAILED DESCRIPTION:
The gap that could noticeably be found in the available literature is that the studies done on SGLT2i were almost tested on people who already using ACEi or ARBs, thus it is unclear whether SGLT2i is used as a first-line instead of ACEi/ARB (If ACEi/ARB are contraindicated or intolerable), to what extent it will be effective in managing DKD compared to the proven effect of ACEi/ARBs alone? Although there is one subgroup analysis in the CANVAS trial to compare the effect of SGLT2 on patients who are on RAS blockers versus those without RAS blockers, the total number of participants who are not on RAS is very small (around 20%) compared to the total number of participants.

the study consists of 2 equal arms, non-inferiority RCT that compares the change in the eGFR rate after one year between the ACEi (enalapril) group versus SGLT2i (empagliflozin) group in 212 men and non-pregnant women with DKD whom age 30-65 years old with UACR above 30mg/g and eGFR ranging from 30-90 ml/min/1.73m2. The study hypothesis is that the mean change of the eGFR in the ACEi group - Mean change of the eGFR in the SGLT2i group is < 5 ml/min/1.73m2 after one year.

Results from this study will add to the current literature examining whether the use of SGLT2i, as a first-line or if ACEi is contraindicated or intolerable, is non-inferior to ACEi in preserving kidney function in DKD patients. Superiority could also be declared if present. Further studies with a longer period of time will be required for comparing the long-term effect of both medications on kidneys.

Rational:

* Based on the ADA/EASD 2019 consensus, SGLT2 inhibitors are recommended in patients with type 2 diabetes in patients with CKD to prevent the progression of CKD (Buse et al.,2019).
* The interpretation of the CANVAS subgroup data is that performance of SGLT2i in patients NOT already on RAS inhibitor is good enough that the two 2 equal arms, non-inferiority would be ethically allowable.
* Since the existing data are insufficient to be analyzed to extract the answer to this question, "Which is better, an ACEI/ARB or an SGLT2i, to delay the progression of renal impairment?" we already know that the combination is effective but some patients may have a choice to make of one OR the other, this study provides a unique opportunity to tackle this gap in the literature.

The reasons beyond the choice of Empagliflozin in this trial were based on many factors. the results of (the EMPA-REG OUTCOME) trial proved its efficacy in delaying the deterioration of kidney function and its availability in the local market. Moreover, it has a good safety profile in comparison to Canagliflozin (ex: risk of bone fracture, lower limb amputation).

ELIGIBILITY:
Inclusion Criteria:

* Men& women with Type 2 Diabetic patient
* Age 30-65 years old
* UACR above 30mg/g
* eGFR between 30-90 ml/min/1.73m2
* Signed and dated informed consent
* Women must agree to use an effective birth control method if they are heterosexually active during the trial and should have a negative pregnancy test on day 1

Exclusion Criteria:

* T1DM, History of diabetic ketoacidosis, beta-cell or pancreas transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Age below 30 and above 65 years old
* hyperkalemia (i.e., K above 6)
* ESRF& e GFR less than 30 ml/min/1.73m2
* renal artery stenosis
* type2 DM pregnant woman & gestational DM, breastfeeding
* history of prior amputation or high risk for amputation (including severe peripheral vascular disease, neuropathy, and diabetic foot ulcers)
* History of one or more severe hypoglycemic episodes within 6 months prior to screening Idiopathic or hereditary angioedema
* allergies, or intolerance to trial medications or their excipients

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
estimated glomerular filtration rate | one year
  eGFR rate (determined by the Modification of Diet in Renal Disease [MDRD] equation) in ml/min/1.73m2

SECONDARY OUTCOMES:
the change in Urine Albumin Creatinine Ratio (UACR) | One year
  UACR (determined at first-morning void by at least 2 of 3 specimens obtained over a 3-to-6-month period) in mg/mmol

OTHER OUTCOMES:
blood pressure | One year
  measured in mmHg
the serum creatinine level | one year
  measured in mg/dL
the rates of clinical events (myocardial infarction, ESRD, congestive heart failure, and stroke) | one year
  if happened during the study

CONTACTS AND LOCATIONS:
Overall Officials: Omar T Elfarargi, Principal Investigator — Primary health care corporation of Qatar

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared after the end of the publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: approximately after 6 months of publication and for 4 years.

REFERENCES:
- [Background] Brenner, B. M., Cooper, M. E., De Zeeuw, D., Keane, W. F., Mitch, W. E., Parving, H. H., ... & Shahinfar, S. 2001.